CLINICAL TRIAL: NCT04509024
Title: Examining the Impact of Non-linguistic Incidental Auditory Category Training on Adult Language Acquisition
Brief Title: Incidental Auditory Category Training for Language Learning
Acronym: IACT
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: In response to the COVID-19 pandemic, the long-term follow-up of participants was dropped from the study protocol as we lacked the time and resources to do so. Methods like eye-tracking were also dropped.
Sponsor: Carnegie Mellon University (Other)
Responsible Party: Principal Investigator, Seth Wiener, Associate Professor, Carnegie Mellon University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 1R03HD099382-01 (NIH)
Record Dates: First submitted 2020-08-06; First posted 2020-08-11 (Actual); Results first posted 2024-07-24 (Actual); Last update posted 2024-07-24 (Actual); Status verified 2024-07

CONDITIONS: Healthy; Language
Keywords: Learning; Speech; Cognition
MeSH Terms: conditions — Language; Speech

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Incidental training (Experimental): Participants undergo novel non-linguistic incidental category learning training.
  Interventions: Behavioral: Incidental training
- Explicit training (Experimental): Participants undergo traditional explicit language learning.
  Interventions: Behavioral: Explicit training
- No training (No Intervention): Participants do not undergo any training.
- Classroom training (Experimental): Participants take part in structured classroom learning.
  Interventions: Behavioral: Classroom training
- Classroom and incidental training (Experimental): Participants take part in structured classroom learning and incidental learning.
  Interventions: Behavioral: Classroom and incidental training
- Classroom and explicit training (Experimental): Participants take part in structured classroom learning and explicit learning.
  Interventions: Behavioral: Classroom and explicit training

INTERVENTIONS:
Behavioral: Incidental training — Training involving non-speech sounds embedded in a video-game.
  Arms: Incidental training
Behavioral: Explicit training — Training involving explicit sound and category information
  Arms: Explicit training
Behavioral: Classroom training — Structured adult classroom language training.
  Arms: Classroom training
Behavioral: Classroom and incidental training — Both classroom and incidental training.
  Arms: Classroom and incidental training
Behavioral: Classroom and explicit training — Both classroom and explicit training.
  Arms: Classroom and explicit training

SUMMARY:
The overarching goal of the proposed research is to understand how human listeners learn speech categories. The project takes a prospective approach with adult second-language learners, blending empirical, methodological and theoretical advances from laboratory studies with explicit classroom instruction. The central hypothesis is that incidentally-acquired nonlinguistic perceptual building block categories may support speech perception and production in a second language. The project will advance important theoretical debates about the cross-talk between general auditory representations and speech categories and will provide a novel approach to nudging adult learners off learning plateau typically encountered in classroom instruction.

DETAILED DESCRIPTION:
Robust speech communication requires that listeners learn linguistically-relevant representations for stable language regularities, such as the speech sounds (phonemes) that convey meaning. In an increasingly multilingual society, as many as twenty percent of Americans accomplish this across multiple languages. Yet, second language acquisition is especially challenging among adult language learners, for whom learning typically involves explicit classroom instruction. Troublingly, research documents that instruction routinely results in a 'learning plateau' whereby language abilities stagnate or even atrophy despite continued instruction. There is a need to establish effective new approaches to nudge adult language learners off this plateau. This project integrates theoretical and methodological developments in auditory category learning with approaches to classroom-based L2 instruction. Specifically, incidental category learning (in which learners' attention is directed away from to-be-learned categories by an engaging videogame) taps into category learning systems distinct from those engaged in more explicit learning. Moreover, incidental learning of nonspeech sound categories leads to activation of putatively speech-selective cortex associated with speech categorization, suggesting potential representational cross-talk. This guides the central hypothesis of the project: incidental learning of nonspeech perceptual building block categories may provide a 'back door' through which to influence adult L2 learners' speech acquisition and to move them off the classroom learning plateau. An intensive 8-week incidental training study will test the hypothesis (Aim 1). Comparison of incidental nonspeech training with explicit L2 speech training will assess whether this cognitive 'back door' may be more effective in promoting L2 speech perception and production than explicit training with L2 speech and will determine the extent to which each interacts with classroom instruction in the L2 (Aim 2). The results will reveal whether nonspeech, auditory categories sharing common perceptual dimensions with second language categories scaffold L2 acquisition, the degree to which explicit instruction may support or interfere with new auditory categories, whether incidental learning is retained after training, and whether learning gains transfer to support other language-learning tasks. In blending empirical, methodological, and theoretical advances from laboratory studies with explicit classroom learning it will be possible to determine the interplay between incidentally-acquired nonlinguistic perceptual building block categories and an emerging L2. This will advance important theoretical debates about the cross-talk between general auditory representations and speech categories and will provide a novel approach to L2 pedagogy.

ELIGIBILITY:
Inclusion Criteria:

* 18 or older, normal hearing
* Native/non-native Chinese speakers

Exclusion Criteria:

* Younger than 18, loss of hearing

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2022-11-01 (Actual); Study Completion 2023-01-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Seth Wiener, PhD, Principal Investigator — Carnegie Mellon University
Locations (1):
- Carnegie Mellon University, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
Participants who have agreed to share their behavioral responses and speech recordings will have their data anonymized and shared via a free, open platform like OpenScience after completion of the study.
Supporting Information: Analytic Code
Time Frame: Anonymized behavioral data available permanently via the Open Science Framework.
Access Criteria: Available via Open Science Framework link
URL: https://osf.io/xjcvg/

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This is the number of participants who agreed to participate in the study following completion of the informed consent process.
Groups:
- Incidental Training: Participants undergo incidental, non-speech training.
- No Training: Participants do not undergo training.
- Classroom Training: Participants undergo structured classroom training.
- Classroom and Incidental Training: Participants undergo both classroom and incidental training.
- Classroom and Explicit Training: Participants undergo both classroom and explicit training.
Period: Overall Study
Arm/Group | Incidental Training | Explicit Training | No Training | Classroom Training | Classroom and Incidental Training | Classroom and Explicit Training
Started | 18 | 17 | 19 | 17 | 18 | 17
Completed | 18 | 17 | 19 | 17 | 18 | 17
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Incidental Training: Participants play a video-game involving non-speech.
- Explicit Training: Participants use a website involving explicit sounds and labels.
- No Training: Participants do not undergo training between pre- and post-tests.
- Classroom Training: Participants take part in a weekly structured language class.
- Classroom and Incidental Training: Participants take part in classroom and video-game training.
- Classroom and Explicit Training: Participants take part in classroom and explicit web-based training.
- Total: Total of all reporting groups
Arm/Group | Incidental Training | Explicit Training | No Training | Classroom Training | Classroom and Incidental Training | Classroom and Explicit Training | Total
Number analyzed (Participants) | 18 | 17 | 19 | 17 | 18 | 17 | 106
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 18 | 17 | 19 | 17 | 18 | 17 | 106
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 20.5 (3.07) | 21.1 (2.37) | 19.8 (2.29) | 20.9 (2.66) | 20.6 (2.40) | 20.6 (3.43) | 20.8 (2.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 11 | 10 | 7 | 11 | 8 | 55
  Male | 10 | 6 | 9 | 10 | 7 | 9 | 51
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 7 | 5 | 6 | 7 | 8 | 7 | 40
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 2 | 1 | 1 | 2 | 1 | 2 | 9
  White | 8 | 9 | 9 | 7 | 7 | 6 | 46
  More than one race | 0 | 1 | 1 | 1 | 2 | 2 | 7
  Unknown or Not Reported | 1 | 1 | 2 | 0 | 0 | 0 | 4
Region of Enrollment [Number; unit: participants]
  United States | 18 | 17 | 19 | 17 | 18 | 17 | 106

OUTCOME MEASURES:

1. Primary Outcome: Change in Sensitivity (D-prime) to Novel Speech Sounds After 2 Months of Training
Description: Each participant's 96 auditory discrimination data points at Pre-test and Post-test, respectively, were reduced to one sensitivity score: d-prime (d': hits minus false alarms). This transformation takes into account response bias and approaches a normal distribution. A higher score represents greater sensitivity. The difference in scores from pre- to post-test represents the change.
Time Frame: Pre-test (baseline) and immediately after 2 months of training.
Measure: Mean (Standard Deviation); unit: sensitivity (d-prime)
Groups:
- Incidental Training: Participants undergo incidental training involving non-speech sounds within a video-game.
- Explicit Training: Participants undergo explicit training involving a website with sound and category labels.
- No Training: Participants did not undergo training between pre- and post-tests.
Arm/Group | Incidental Training | Explicit Training | No Training | Classroom Training | Classroom and Incidental Training | Classroom and Explicit Training
Number analyzed (Participants) | 18 | 17 | 19 | 17 | 18 | 17
sensitivity (d-prime) | 1.51 (1.36) | 0.47 (1.51) | 0.53 (.96) | 1.33 (1.68) | 1.33 (1.32) | 1.23 (1.12)

2. Primary Outcome: Change in Auditory Category Learning Accuracy After 2 Months of Training
Description: Each participant's 96 auditory categorization data points at Pre-test and Post-test, respectively, were turned into a mean of the correct answers. The difference between the two accuracy scores represents the mean change in accuracy.
Time Frame: Pre-test (baseline) and immediately after 2 months of training.
Measure: Mean (Standard Deviation); unit: percentage of correct trials
Arm/Group | Incidental Training | Explicit Training | No Training | Classroom Training | Classroom and Incidental Training | Classroom and Explicit Training
Number analyzed (Participants) | 18 | 17 | 19 | 17 | 18 | 17
percentage of correct trials | .43 (.19) | .31 (.26) | .04 (.11) | .48 (.2) | .44 (.13) | .49 (.21)

3. Primary Outcome: Novel Auditory Word Learning Accuracy After 2 Months of Training
Description: At post-test, participants did a three day novel word learning task. Their 48 word identification data points on the first and third days, respectively, were turned into a mean correct score. The difference in scores from Day 1 to Day 3 represents the change in mean novel word learning accuracy.
Time Frame: Immediately after 2 months of training.
Measure: Mean (Standard Deviation); unit: percentage of correct trials
Arm/Group | Incidental Training | Explicit Training | No Training | Classroom Training | Classroom and Incidental Training | Classroom and Explicit Training
Number analyzed (Participants) | 18 | 17 | 19 | 17 | 18 | 17
percentage of correct trials | .06 (.24) | 0 (.12) | -.03 (.16) | -.04 (.13) | .1 (.2) | .09 (.12)

4. Secondary Outcome: Word Recognition Accuracy in Unrelated Language 3 Months After Training
Description: Three months after training, participants were scheduled to learn words in an unrelated language. Their mean accuracy would be calculated.
Time Frame: 3 months post-intervention
Population: This component of the project was cancelled due to the COVID-19 pandemic and no data were collected.
Arm/Group | Incidental Training | Explicit Training | No Training | Classroom Training | Classroom and Incidental Training | Classroom and Explicit Training
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Participants were monitored and assessed for three months.
Description: Participants were tested in-person or via web-cam.
  Participants at risk for Serious Adverse Events was 106. Participants at risk for All-Cause Mortality was 106.
  Participants at risk for Other (Not Including Serious) Adverse Events was 106.
Arm/Group | Incidental Training | Explicit Training | No Training | Classroom Training | Classroom and Incidental Training | Classroom and Explicit Training
All-Cause Mortality (participants affected / at risk) | 0/18 | 0/17 | 0/19 | 0/17 | 0/18 | 0/17
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/17 | 0/19 | 0/17 | 0/18 | 0/17
Other Adverse Events (participants affected / at risk) | 0/18 | 0/17 | 0/19 | 0/17 | 0/18 | 0/17

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-02-26): https://cdn.clinicaltrials.gov/large-docs/24/NCT04509024/Prot_SAP_001.pdf
  • Informed Consent Form (2021-06-05): https://cdn.clinicaltrials.gov/large-docs/24/NCT04509024/ICF_002.pdf